CLINICAL TRIAL: NCT03054064
Title: Evaluating the Indego Exoskeleton for Persons With Hemiplegia Due to CVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Hannifin Corporation (Industry)
Collaborators: Shepherd Center, Atlanta GA (Other); Cedars-Sinai Medical Center (Other); Sheltering Arms Physical Rehabilitation Hospitals (Other); Shirley Ryan AbilityLab (Other); Kessler Foundation (Other); St. Charles Hospital (Unknown); TIRR Memorial Hermann (Other); Rusk Rehabilitation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHIND_CVA01
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Cerebrovascular Accident (CVA); Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All Enrolled Subjects (Experimental): All enrolled subjects will receive gait training with the Indego.
  Interventions: Device: Indego Exoskeleton

INTERVENTIONS:
Device: Indego Exoskeleton — Six study sessions including five Indego training sessions over two weeks.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Indego exoskeleton as a gait training tool for individuals with hemiplegia due to Cerebrovascular Accident (CVA).

ELIGIBILITY:
Inclusion Criteria:

* Height 5'1" to 6'3" (acceptable height may vary by a few inches depending on femur length)
* Weight 250 pounds or less
* History of one sided ischemic or hemorrhagic stroke with resultant hemiparesis
* Manual Muscle Test (MMT) 4/5 in at least upper extremity
* No restrictions on time since stroke (acuity), but all subjects need to be cleared by MD for locomotor training
* No other brain abnormalities or neurological diseases/disorders
* Has not been diagnosed with more than one stroke
* Passive range of motion (PROM) at shoulders, trunk, hips, knees and ankles within functional limits for safe gait
* Skin intact where interfaces with Indego device
* Modified Ashworth Scale (MAS) for spasticity 3 or less in the lower extremities
* Absence of complicating physical or mental conditions as determined by MD that would preclude the individual from safely participating in gait training
* Must be able to follow directions and communicate basic needs, demonstrated by a Mini- Mental State Exam (MMSE) score of 18 or greater

Exclusion Criteria:

* Failure to meet all inclusion criteria
* Pregnancy
* Colostomy bag
* Uncontrolled/untreated hyper- or hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cedars-Sinai Health System, Los Angeles, California
  - Shepherd Center, Atlanta, Georgia
  - Rehabilitation Institute of Chicago (Shirley Ryan AbilityLab), Chicago, Illinois
  - Kessler Foundation, West Orange, New Jersey
  - St. Charles Hospital, Port Jefferson, New York
  - TIRR Memorial Hermann, Houston, Texas
  - Sheltering Arms Physical Rehabilitation Centers, Mechanicsville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 48
Screen Failure | 2
Completed | 42
Not Completed | 6
Not completed — Lower Extremity Deep Vein Thrombosis | 1
Not completed — Investigator Decision | 2
Not completed — Bladder Issue | 1
Not completed — High Blood Pressure | 1
Not completed — Change in Status | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3
  Race: Black or African American | 7
  Race: White | 25
  Race: Hispanic, Latino or other Spanish origin | 7
Acuity of Cerebrovascular Accident (CVA) [Count of Participants; unit: Participants] — Acute: less than 2 months since CVA, Sub-acute: 2-6 months since CVA, or Chronic: more than 6 months since CVA
  Participants
    Acute | 3
    Subacute | 6
    Chronic | 33
Severity of Cerebrovascular Accident (CVA) [Count of Participants; unit: Participants] — Mild: Fugl-Meyer Motor Assessment score greater than 79, Moderate: Fugl-Meyer Motor Assessment score 56-79, Severe: Fugl-Meyer Motor Assessment score 36-55, or Very Severe: Fugl-Meyer Motor Assessment score 0-35
  Participants
    Mild | 4
    Moderate | 10
    Severe | 15
    Very Severe | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety of Individuals With Hemiplegia Due to CVA Using the Indego Measured Through Reported Subject Adverse Events and Serious Adverse Events
Description: Safety of individuals with hemiplegia due to CVA using the Indego measured through reported Subject Adverse Events and Serious Adverse Events
Time Frame: 2 weeks
Measure: Number; unit: Events
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 42
Events
  Trial-related Adverse Events | 3
  Trial-related Serious Adverse Events | 0

2. Secondary Outcome: Spasticity of Bilateral Upper Extremities (UE) and Lower Extremities (LE) Measured With Modified Ashworth Scale
Description: Spasticity measured with Modified Ashworth Scale (MAS)
  0 - No increase in muscle tone
  1 - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM) 2 - More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved 3 - Considerable increase in muscle tone, passive movement difficult 4 - Affected part(s) rigid in flexion or extension
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 42
units on a scale
  Average MAS Right UE Session 1 | 1 (1.4)
  Average MAS Left UE Session 1 | 1 (1.5)
  Average MAS Right LE Session 1 | 1 (1.1)
  Average MAS Left LE Session 1 | 1 (1.2)
  Average MAS Right UE Session 6 | 1 (1.4)
  Average MAS Left UE Session 6 | 1 (1.3)
  Average MAS Right LE Session 6 | 1 (1.0)
  Average MAS Left LE Session 6 | 1 (1.1)

3. Secondary Outcome: Activity Measured by Functional Ambulation Category
Description: Activity measured by Functional Ambulation Category (FAC)
  1. unable to ambulate/ambulates only in parallel bars/requires supervision or physical assistance from > 1 person
  2. requires manual contact of one person during ambulation on level surfaces/manual contact is continuous and necessary to support body weight and/or to maintain balance or assist coordination
  3. requires manual contact of one person during ambulation on level surfaces/manual contact is continuous or intermittent light touch to assist balance or coordination
  4. ambulation occurs on level surfaces without manual contact of another person/requires stand-by guarding of one person because of poor judgment, questionable cardiac status, or the need for verbal cuing to complete the task
  5. ambulation is independent on level surfaces/requires supervision/physical assistance to negotiate stairs, inclines, or unlevel surfaces
  6. ambulation is independent on unlevel and level surfaces, stairs and inclines
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 42
units on a scale
  Average FAC Session 1 | 5 (2)
  Average FAC Session 6 | 5 (1)

4. Secondary Outcome: Gait Speed (Without Indego) Measured With 10 Meter Walk Test
Description: 10 Meter Walk Test (MWT) without Indego to measure gait speed
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 42
seconds
  Average 10 MWT time Session 1 | 24.4 (20.4)
  Average 10 MWT time Session 6 | 19.4 (12.9)

5. Secondary Outcome: Pain Measured With Face, Legs, Activity, Cry, Consolability Scale
Description: Pain measured with Face, Legs, Activity, Cry, Consolability (FLACC) Scale Face 0: no particular expression or smile
  1. occasional grimace or frown, withdrawn, disinterested
  2. frequent to constant frown, clenched jaw, quivering chin
  Legs 0: normal position or relaxed
  1. uneasy, restless, tense
  2. kicking, or legs drawn up
  Activity 0: lying quietly, normal position, moves easily
  1. squirming, shifting back and forth, tense
  2. arched, rigid, or jerking
  Cry 0: no cry (awake or asleep)
  1. moans or whimpers, occasional complaint
  2. crying steadily, screams or sobs, frequent complaints
  Consolability 0: content, relaxed
  1. reassured by occasional touching, hugging, or being talked to, distractable
  2. difficult to console or comfort
  Minimum score: 0 Maximum Score: 10
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 42
units on a scale
  Average FLACC Session 1 | 0 (0)
  Average FLACC Session 6 | 0 (0)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 3/48
Other Adverse Events (participants affected / at risk) | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=48)
Urinary Retention (Renal and urinary disorders) | 1 (1) — Patient was admitted to hospital for urinary retention that was resolved with foley catheter. Adverse Event determined to be unrelated to study and device.Subject withdrew from study.
High blood pressure (General disorders) | 1 (1) — Patient came to first Indego session and had BP 180/125. Patient admitted to hospital and they indicated that they forgot to take their BP medication that morning. Adverse Event determined to be unrelated to study/device. Subject withdrew from study.
Deep vein thrombosis (General disorders) | 1 (1) — Patient was admitted to hospital for lower extremity deep vein thrombosis after being consented for study but before beginning first session. Adverse Event determined to be unrelated to study and device. Subject withdrew from study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Subjects (N=48)
Loss of balance (Product Issues) | 1
Pain (Musculoskeletal and connective tissue disorders) | 1
Abrasion (Skin and subcutaneous tissue disorders) | 1
Fall (General disorders) | 1 — Patient noted posterior loss of balance falling after attempting to retrieve pillow off ground at home while gripping walker. Determined to be unrelated to study and device.
Abrasion (Skin and subcutaneous tissue disorders) | 1 — Subject had skin abrasion from personal AFO use on left lateral calf. Area did not come in contact with Indego and was present prior to use.
Abrasion (Skin and subcutaneous tissue disorders) | 1 — Additional areas of breakdown and blisters from subject's personal AFO developed over the weekend (between Indego sessions).
Fall (General disorders) | 1 — Patient reported fall out of wheelchair. Determined to be unrelated to study and device.
Change in status (General disorders) | 1 — Patient had been consented for study but upon arriving for first session subject had poor verbal responsiveness with increased pushing behavior. Change in status determined to be unrelated to study and device. Subject withdrew from study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT03054064/Prot_SAP_000.pdf